CLINICAL TRIAL: NCT01727674
Title: Exploring the Experience of Communication for Patients With Depression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207022RIB
Record Dates: First submitted 2012-11-02; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Depression
Keywords: Depression; experiences of communication
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
According to the statistics released by the Department of Health,Executive Yuan in 2005,depression, cancer and AIDS will become the three main diseases of the 21st century.The prevalence of depression is 5.8% for males and 9.5% for women in the worldwide total population each year.Depression ranks second next to cardiovascular disease and impacts on social and economic burdens.From the perspectives of prevalence,suicide rate,loss of workforce,family burden,co-morbidities and health care expenses,the issues related to caring for patients with depression should not be overlooked.Communication is often neglected while exploring the issues of caring for depressed patients,which can consequently affect their family,work performance,social interaction,and even leads to a risk of suicide.Therefore,in order to enhance their psychological adjustment and health management,it is particularly important to achieve effective communications.

DETAILED DESCRIPTION:
This study aims to investigate the experiences of communication for patients with depression.Purposive sampling will be used to recruit participants in this study.Eligible participants consist of those who attend the outpatient department of psychiatry regularly,have emotional stability and clear consciousness,More than 20 years old,can be communicated in Mandarin or Taiwanese,and are willing to take the interviews.In-depth interviews will be conducted to collect qualitative data,and data will be categorized and analyzed according to Tesch(1990).Sampling will be stopped until data saturation.The findings may be referenced by the relevant agencies and medical institutions to care the patients with depression,as well as provide a basis for nursing care and education.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric physician-diagnosed patients with major depression,including major depressive disorder,identified patients with stable and stable condition treatment by a physician.
* Able to communicate to the language of the country or Taiwan.
* by explanations can share experiences,and has executed a written consent to.

Exclusion Criteria:

* Combined with other mental illness.
* Depression in patients with unstable condition,including serious and has a tendency to suicide,violence and attacks.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: depression
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Exploring the experience of communication for patients with depression | six months
  * The study does not involve drugs or invasive test.
  * Does not have hurt the lives of the respondents.
  * Your information anonymous and efforts to provide 24-hour contact line and other mechanisms,the inconvenience or injury to reduce.

CONTACTS AND LOCATIONS:
Overall Officials: Jui-Ching Hong, MASTER, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Hsinchu, Taiwan